CLINICAL TRIAL: NCT03969420
Title: A Phase 2, Open-label, Randomized, Two-stage Clinical Study of Alvocidib in Patients With Relapsed/Refractory Acute Myeloid Leukemia Following Treatment With Venetoclax Combination Therapy
Brief Title: Study of Alvocidib in Patients With Relapsed/Refractory AML Following Treatment With Venetoclax Combination Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision to terminate the development of alvocidib program on 17 November 2020. Patients permitted on treatment until April 22, 2021. The last end-of-treatment follow-up completed on May 14, 2021.
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TPI-ALV-202
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Results first posted 2022-10-19 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Tolero, Phase 2, AML, Relapsed, Refractory, Alvocidib, Venetoclax
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — alvocidib; Cytarabine

STUDY DESIGN:
Intervention Model Description: Randomized, Two-stage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Lead-In Cohort: Arm 1 (Experimental): Refractory (i.e., failed to achieve a CR/CRi or achieved a CR/CRi with duration <90 days)
  Interventions: Drug: Alvocidib (flavopiridol) and cytarabine (Ara-C)
- Lead-In Cohort: Arm 2 (Experimental): Relapsed (i.e., reoccurrence of disease following a CR/CRi with duration ≥90 days).
  Interventions: Drug: Alvocidib (flavopiridol)
- Stage 1: Arm 1 (Experimental): Refractory (i.e., failed to achieve a CR/CRi or achieved a CR/CRi with duration <90 days)
  Interventions: Drug: Alvocidib (flavopiridol) and cytarabine (Ara-C)
- Stage 1: Arm 2 (Experimental): Relapsed (i.e., reoccurrence of disease following a CR/CRi with duration ≥90 days).
  Interventions: Drug: Alvocidib (flavopiridol)

INTERVENTIONS:
Drug: Alvocidib (flavopiridol) and cytarabine (Ara-C) — Alvocidib (flavopiridol), administered intravenously, + cytarabine (Ara-C), administered by subcutaneous injection
  Arms: Lead-In Cohort: Arm 1; Stage 1: Arm 1
Drug: Alvocidib (flavopiridol) — Administered intravenously
  Arms: Lead-In Cohort: Arm 2; Stage 1: Arm 2

SUMMARY:
This study will evaluate the safety and efficacy of alvocidib in patients with AML who have either relapsed from or are refractory to venetoclax in combination with azacytidine or decitabine.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥18 years of age.
2. Have an established, pathologically confirmed diagnosis of AML by World Health Organization (WHO) criteria, excluding acute promyelocytic leukemia (APL-M3) with a bone marrow of >5% blasts based on histology or flow cytometry.
3. Have received initial induction therapy with venetoclax in combination with azacytidine or decitabine (with or without other investigational agents as part of a clinical trial; requires Medical Monitor review) and were either refractory (failed to achieve a CR/CRi or achieved a CR/CRi with duration <90 days) or have relapsed (reoccurrence of disease following a CR/CRi with duration ≥90 days).
4. Have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤2.
5. Have a glomerular filtration rate (GFR) ≥30 mL/min using the Cockcroft-Gault equation.
6. Have an alanine aminotransferase (ALT)/aspartate aminotransferase (AST) level ≤5 times upper limit of normal (ULN).
7. Have a total bilirubin level ≤2.0 mg/dL (unless secondary to Gilbert syndrome, hemolysis, or leukemia).
8. Be infertile or agree to use an adequate method of contraception:sexually active patients and their partners must use an effective method of contraception associated with a low failure rate prior to study entry, for the duration of study participation, and for at least 3 months (males) and 6 months (females) after the last dose of study drug.
9. Be able to comply with the requirements of the entire study.
10. Provide written informed consent prior to any study related procedure: in the event that the patient is re-screened for study participation or a protocol amendment alters the care of an ongoing patient, a new informed consent form must be signed.

Exclusion Criteria:

1. Received any previous treatment with alvocidib or any other CDK inhibitor or received prior anti-leukemic therapy other than first-line venetoclax in combination with azacytidine or decitabine.
2. Require concomitant chemotherapy, radiation therapy, or immunotherapy. Hydroxyurea is allowed up to the evening before starting (but not within 12 hours) of starting treatment on either arm.
3. Received an allogeneic stem cell transplant within 60 days of the start of study treatment. Patients who received an allogeneic stem cell transplant must be off all immunosuppressants at the time of study treatment
4. Are receiving or have received systemic therapy for graft-versus-host disease.
5. Have a peripheral blast count of >30,000/mm3 (may use hydroxyurea as in #2 above).
6. Received antileukemic therapy within the last 2 weeks or 3-5 half lives of the prior therapy (with the exception of hydroxyurea or if the patient has definite refractory disease), whichever is less. Refractory patients who received therapy within the last 2 weeks may be eligible with prior approval of the Medical Monitor.
7. Diagnosed with acute promyelocytic leukemia (APL-M3).
8. Have active central nervous system (CNS) leukemia.
9. Have evidence of uncontrolled disseminated intravascular coagulation.
10. Have an active, uncontrolled infection.
11. Have other life-threatening illness.
12. Have other active malignancies requiring treatment or diagnosed with other malignancies within the last 6 months, except nonmelanoma skin cancer or cervical intraepithelial neoplasia.
13. Have mental deficits and/or psychiatric history that may compromise the ability to give written informed consent or to comply with the study protocol.
14. Are pregnant and/or nursing.
15. Have received any live vaccine within 14 days prior to first study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2021-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Anthony, DO, Study Director — Sumitomo Pharma America, Inc.
Locations (18):
- United States (18):
  - Community Medical Providers, Clovis, California
  - City of Hope National Medical Center, City of Hope Medical Center, Duarte, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - University of California, San Francisco Medical Center, San Francisco, California
  - Advent Health Medical Group Blood & Marrow Transplant at Orlando, Orlando, Florida
  - Orlando Health, Inc, Univ of Florida Health Cancer Center, Orlando, Florida
  - Indiana Blood and Marrow Translplantation - Clinic, Indianapolis, Indiana
  - University of Kansas Medical Center, Westwood, Kansas
  - Ochsner Medical Center, New Orleans, Louisiana
  - University of New Mexico, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - University of North Carolina (UNC), Chapel Hill, North Carolina
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Sciences University - Knight Cancer Institute - Center for Hematologic Malignancies, Portland, Oregon
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Baylor University Center, Dallas, Texas
  - University of Washington, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eleven subjects were enrolled between January 2020 and November 2020
Pre-assignment Details: A safety lead-in cohort comprised of 6 patients (3 patients in each treatment arm) were treated and evaluated for dose-limiting toxicities (DLTs) prior to enrolling patients in Stage 1. (Seven patients were enrolled but only 6 were considered evaluable.) If a DLT was observed, dose de-escalation occurred, and if no DLTs were observed, randomization into Stage 1 would commence.
Groups:
- Lead-In Cohort: Arm 1; Stage 1: Arm 1: ALDAC: Alvocidib administered intravenously on days 1 and 15 + cytarabine administered by subcutaneous injection days 3-12 of each 28 day cycle. Patients were stratified based on response to prior therapy (i.e. Refractory or Relapsed)
- Lead-In Cohort: Arm 2; Stage 1: Arm 2: ALV: Alvocidib administered intravenously on days 1, 8 and 15 of each 28 day cycle. Patients were stratified based on response to prior therapy (i.e. Refractory or Relapsed)
Period: Overall Study
Arm/Group | Lead-In Cohort: Arm 1 | Lead-In Cohort: Arm 2 | Stage 1: Arm 1 | Stage 1: Arm 2
Started | 3 (Any patient who received at least 1 dose of study drug) | 4 (Any patient who received at least 1 dose of study drug) | 2 (Any patient who received at least 1 dose of study drug) | 2 (Any patient who received at least 1 dose of study drug)
Completed | 3 (Any patient who received at least 1 dose of study drug) | 4 (Any patient who received at least 1 dose of study drug) | 2 (Any patient who received at least 1 dose of study drug) | 2 (Any patient who received at least 1 dose of study drug)
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lead-In Cohort: Arm 1 | Lead-In Cohort: Arm 2 | Stage 1: Arm 1 | Stage 1: Arm 2 | Total
Number analyzed (Participants) | 3 | 4 | 2 | 2 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 1 | 1 | 2
  >=65 years | 3 | 4 | 1 | 1 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 1 | 6
  Male | 1 | 2 | 1 | 1 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 3 | 2 | 2 | 9
  Black | 1 | 0 | 0 | 0 | 1
  Hispanic | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0 | 0
  Not reported | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Combined Complete Remission
Description: Rate of combined complete remission (complete remission (CR) + CR with incomplete hematological recovery (CRi)), as defined by the International Working Group Criteria and 2017 European LeukemiaNet).
  Combined complete remissions (patients with a best response of CR or CRi), complete remissions, composite complete remissions (patients with a best response of CR, CRi or CRh), and combined responses (patients with a best response of CR, CRi, CRh, MLFS or PR) will be summarized by observed response rates and estimated 95% CIs.
Time Frame: Response assessments were measured from date of first dose through End of Treatment date, an average of 3 months.
Population: The sponsor decided not to continue the study based on the overall company strategy in AML. Data collection and analysis were not conducted.
Arm/Group | Lead-In Cohort: Arm 1 | Lead-In Cohort: Arm 2 | Stage 1: Arm 1 | Stage 1: Arm 2
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Median Overall Survival
Description: Time from treatment (Day 1) until death from any cause
Time Frame: From first dose until disease progression or death; through study termination, an average of 10 months
Population: as for outcome 1
Arm/Group | Lead-In Cohort: Arm 1 | Lead-In Cohort: Arm 2 | Stage 1: Arm 1 | Stage 1: Arm 2
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Complete Response Rate
Description: Percentage of patients achieving complete response (CR) whose bone marrow is determined to be negative for minimal residual disease (MRD) using standardized techniques (ie, multiparametric flow cytometry [MPFC] and molecular testing including next generation sequencing [NGS]
Time Frame: Response assessments were measured from date of first dose through end of treatment date, an average of 3 months
Population: as for outcome 1
Arm/Group | Lead-In Cohort: Arm 1 | Lead-In Cohort: Arm 2 | Stage 1: Arm 1 | Stage 1: Arm 2
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Composite CR Rate
Description: Patients with a best response of CR + CRi + CRh (CR + partial recovery of both blood cell types)
Time Frame: Response assessments were measured from date of first dose through end of treatment date, an average of 3 months
Population: as for outcome 1
Arm/Group | Lead-In Cohort: Arm 1 | Lead-In Cohort: Arm 2 | Stage 1: Arm 1 | Stage 1: Arm 2
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Combined Response Rate
Description: Combined Percentage of Patients Achieving One of the Following: CR < CRi, CRh, MLFS, PR
  Morphologic leukemia-free state (MLFS) = Bone marrow blasts <5%; absence of blasts with Auer rods; absence of extramedullary disease; no hematologic recovery required;
  Partial Response (PR) = Meets all hematologic values required for CR but with a decrease of at least 50% in the percentage of blasts to ≥5% to ≤25% in bone marrow
Time Frame: Response assessments were measured from date of first dose through end of treatment date, an average of 3 months
Population: as for outcome 1
Arm/Group | Lead-In Cohort: Arm 1 | Lead-In Cohort: Arm 2 | Stage 1: Arm 1 | Stage 1: Arm 2
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Event Free Survival (EFS)
Description: Event Free Survival - time from first treatment (D1) until (a) treatment failure, (b) relapse after CR/Cri or CRh, or (c) death from any cause, whichever occurs first
Time Frame: From first dose until disease progression or death; through study termination, an average of 10 months
Population: as for outcome 1
Arm/Group | Lead-In Cohort: Arm 1 | Lead-In Cohort: Arm 2 | Stage 1: Arm 1 | Stage 1: Arm 2
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Duration of Composite Complete Remission (CR)
Description: Duration of Composite CR, defined as the time from first documented response of CR, CRi or CRhi to relapse or death from any cause
Time Frame: Response assessments were measured from date of first dose through end of treatment date, an average of 3 months
Population: as for outcome 1
Arm/Group | Lead-In Cohort: Arm 1 | Lead-In Cohort: Arm 2 | Stage 1: Arm 1 | Stage 1: Arm 2
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Transfusion Independence
Description: Rates of 28- and 56-day Transfusion Independence (TI) = Percentages of patients who do not receive red blood cell (RBC) transfusions, platelet (PLT) transfusions, and neither RBC nor PLT transfusions for 28 and 56 days; comprised of 6 secondary endpoints
Time Frame: Transfusion dependence was measured from 28 days prior to first dose through 56 days after last dose, an average of 6 months
Population: as for outcome 1
Arm/Group | Lead-In Cohort: Arm 1 | Lead-In Cohort: Arm 2 | Stage 1: Arm 1 | Stage 1: Arm 2
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious and Other Adverse Events were assessed from the date of first treatment through 30 days of the last administration of study drug, an average of 4 months. All-Cause Mortality was assessed from the date of first treatment until death, up to 14 months.
Arm/Group | Lead-In Cohort: Arm 1 | Lead-In Cohort: Arm 2 | Stage 1: Arm 1 | Stage 1: Arm 2
All-Cause Mortality (participants affected / at risk) | 2/3 | 3/4 | 1/2 | 1/2
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/4 | 2/2 | 1/2
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lead-In Cohort: Arm 1 (N=3) | Lead-In Cohort: Arm 2 (N=4) | Stage 1: Arm 1 (N=2) | Stage 1: Arm 2 (N=2)
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0 | 0
Corona virus infection (Infections and infestations) | 0 | 0 | 1 | 0
sepsis (Infections and infestations) | 0 | 1 | 0 | 0
disease progression (General disorders) | 0 | 1 | 1 | 0
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Acute myeloid leukaemia refractory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lead-In Cohort: Arm 1 (N=3) | Lead-In Cohort: Arm 2 (N=4) | Stage 1: Arm 1 (N=2) | Stage 1: Arm 2 (N=2)
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 1 | 0
nausea (Gastrointestinal disorders) | 0 | 1 | 2 | 1
vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0
abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0
stomatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2 | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 1 | 0
sepsis (Infections and infestations) | 0 | 2 | 0 | 0
Abscess intestinal (Infections and infestations) | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0 | 0
Corona virus infection (Infections and infestations) | 0 | 0 | 1 | 0
Diverticultits (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 2 | 2 | 0 | 1
Platelet count decreased (Investigations) | 0 | 2 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Blood lactate dehydrogenase (Investigations) | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Disease progression (General disorders) | 0 | 1 | 1 | 0
Catheter site pain (General disorders) | 0 | 1 | 0 | 0
Face oedema (General disorders) | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Acute myeloid leukaemia refractory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/20/NCT03969420/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/20/NCT03969420/SAP_001.pdf